CLINICAL TRIAL: NCT05153967
Title: U01 Cooperative Assessment of Late Effects for Sickle Cell Disease Curative Therapies
Brief Title: Cooperative Assessment of Late Effects for SCD Curative Therapies
Acronym: COALESCE
Status: Recruiting | Type: Observational
Sponsor: Vanderbilt University Medical Center (Other)
Collaborators: Johns Hopkins University (Other); Children's National Research Institute (Other); Emory University (Other); University of Illinois at Chicago (Other); Children's Healthcare of Atlanta (Other)
Responsible Party: Principal Investigator, Michael DeBaun, Professor of Pediatrics and Medicine, Vanderbilt University Medical Center
Other Study IDs: 210806
Record Dates: First submitted 2021-10-25; First posted 2021-12-10 (Actual); Last update posted 2026-01-30 (Actual); Status verified 2026-01

CONDITIONS: Sickle Cell Disease; Pulmonary Disease; Renal Disease; Heart Disease
Keywords: Myeloablative Autologous Gene Editing; Myeloablative Autologous Gene Therapy; Myeloablative allo-HSCT; Nonmyeloablative allo-HSCT; Disease-Modifying Therapy
MeSH Terms: conditions — Anemia, Sickle Cell; Lung Diseases; Kidney Diseases; Heart Diseases

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Other
Biospecimen Retention: Samples With DNA — Blood samples for genetic testing to identify whether genes may predict health outcomes.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (4):
- Pediatric Myeloablative allo-HSCT: Participants ages 4 to 17 years old with SCD who underwent or are scheduled to undergo myeloablative allo-HSCT.
- Pediatric Standard Disease-Modifying Therapy: Participants ages 4 to 17 years old with SCD who receive standard therapy.
- Adult Non-Myeloablative allo-HSCT: Participants ages 18 to 65 years old with SCD who underwent or are scheduled to undergo non-myeloablative allo-HSCT.
- Adult Standard Disease-Modifying Therapy: Participants ages 18 to 65 years old with SCD who receive standard therapy.

SUMMARY:
Sickle Cell Disease is one of the most common genetic diseases in the United States, occurring in approximately 1 in 400 births. Approximately 100,000 individuals are diagnosed with SCD in the United States. Mortality for children with SCD has decreased substantially over the past 4 decades, with >99% of those born in high resource settings, including the United States, France, and England, now surviving to 18 years of age. However, the life expectancy of adults with SCD is severely shortened. Dysfunction of the heart, lung, and kidney is directly associated with decreased life expectancy. With the variety of curative therapies that are now available for SCD, long-term health outcomes studies are time-sensitive. As of now, efforts to determine long-term health outcomes following curative therapies for SCD have been limited. Though curative therapies initially should provide a cure for symptoms of SCD, there is the risk of late health outcomes to consider. Defining health outcomes following curative therapy is essential to improve personalized decision-making when considering curative versus disease-modifying therapeutic options. The primary goal of this study is to determine whether curative therapies for individuals with SCD will result in improved or worsening heart, lung, and kidney damage when compared to individuals with SCD receiving standard therapy. The investigators will also explore whether certain genes are associated with a good or bad outcome after curative therapy for SCD.

DETAILED DESCRIPTION:
Our primary objective is initiating a personalized approach to curative therapies in children and adults with sickle cell disease (SCD) to maximize benefits and limit adverse outcomes. Limited clinical studies exist to determine the long-term health outcomes following curative therapies for SCD. With emerging curative therapies for SCD (allogeneic [allo] hematopoietic stem cell transplant [HSCT], gene therapy/editing), long-term health outcomes studies are critical to inform personalized choices. Unfortunately, adverse outcomes have started to emerge after SCD curative therapy. Thus, risks of a cure in SCD must be measured against the benefits of a cure, including stabilization of lung function (FEV1) and improved tricuspid regurgitant jet velocity [TRJV]. Ultimately, the shortened lifespan of individuals with SCD, attributable to declining heart (elevated TRJV), lung (decreased FEV1), and kidney (decreased eGFR) function, for which curative therapies were designed to ameliorate, must be measured against favorable and unfavorable late outcomes. In our multicenter retrospective-prospective cohort, the investigators will test the following hypotheses: 1a): myeloablative curative therapies for children with SCD will result in progressive pulmonary and renal dysfunction when compared to children with SCD receiving standard therapy; 1b): nonmyeloablative HSCT for adults with SCD will result in no significant change in FEV1% predicted, but will lead to accelerated decline in eGFR when compared to adults receiving standard therapy; 2) nonmyeloablative HSCT for adults with SCD will be associated with a clinically significant improvement in TRJV following HSCT; and 3) in adults with SCD, proliferative and genotoxic stress uniformly related to nonmyeloablative allo-HSCT and myeloablative gene editing will lead to post-HSCT therapy-related myeloid neoplasm of recipient origin. The investigators will address these hypotheses with the following aims: 1) evaluate the incidence of pulmonary and renal function in 1a: children with SCD receiving myeloablative curative therapies; and 1b: adults with SCD receiving nonmyeloablative allo-HSCT, compared to a pre-existing cohort of children and adults with SCD; 2) determine whether there is a clinically significant improvement in TRJV in adults with SCD, at least half having TRJV > 2.5 m/s, following nonmyeloablative allo-HSCT, 3) evaluate the prevalence, incidence and evolution of Clonal hematopoiesis of indeterminate potential (CHIP) concerning therapy-related myeloid neoplasm development following non-myeloablative HSCT or myeloablative gene editing in adults and children with SCD, and 4) evaluate accuracy and gaps involved in collecting clinical health record data directly from patients and family members in comparison to clinical health record data collected by research coordinators.

ELIGIBILITY:
Inclusion Criteria

* Confirmed laboratory diagnosis of SCD
* Ability to give informed consent
* Ability to provide pre- and post-curative therapy data
* Treated with either one HSCT or with standard disease-modifying therapy

Exclusion Criteria

•History of non-compliance

Ages: 4 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Participants will be patient volunteers from the sickle cell disease clinics and transplant centers of participating study sites.
Sampling Method: Non-Probability Sample
Enrollment: 750 (Estimated)
Dates: Start 2022-07-12 (Actual); Primary Completion 2026-06 (Estimated); Study Completion 2027-02 (Estimated)

PRIMARY OUTCOMES:
Measurement of longitudinal change in FEV1 | Through study completion, an average of four years
  Measurements of forced expiratory volume in 1 second (FEV1) based on the global lung index will be acquired from children with SCD receiving myeloablative curative therapies and adults with SCD receiving nonmyeloablative allo-HSCT, as well as from the respective control children and adult cohorts with SCD who received standard therapy. FEV1 will be reported in liters. (References: Eur Respir J. Volume 40 Issue 6: pages 1324-1343, 2012 June 27; Am J Hematol. Volume 93 Issue 3: pages 408-415, 2018 March).
Percent predicted value of longitudinal change in FEV1 | Through study completion, an average of four years
  Percent predicted of forced expiratory volume in 1 second (FEV1) based on the global lung index will be acquired from children with SCD receiving myeloablative curative therapies and adults with SCD receiving nonmyeloablative allo-HSCT, as well as from the respective control children and adult cohorts with SCD who received standard therapy. FEV1 will be reported in percentage. (References: Eur Respir J. Volume 40 Issue 6: pages 1324-1343, 2012 June 27; Am J Hematol. Volume 93 Issue 3: pages 408-415, 2018 March).
Measurement of longitudinal change in FVC | Through study completion, an average of four years
  Measurements of forced volume capacity (FVC) based on the global lung index will be acquired from children with SCD receiving myeloablative curative therapies and adults with SCD receiving nonmyeloablative allo-HSCT, as well as from the respective control children and adult cohorts with SCD who received standard therapy. FVC will be reported in liters. (References: Eur Respir J. Volume 40 Issue 6: pages 1324-1343, 2012 June 27; Am J Hematol. Volume 93 Issue 3: pages 408-415, 2018 March).
Percent predicted value of longitudinal change in FVC | Through study completion, an average of four years
  Percent predicted of forced volume capacity (FVC) on the global lung index will be acquired from children with SCD receiving myeloablative curative therapies and adults with SCD receiving nonmyeloablative allo-HSCT, as well as from the respective control children and adult cohorts with SCD who received standard therapy. FVC will be reported in percentage. (References: Eur Respir J. Volume 40 Issue 6: pages 1324-1343, 2012 June 27; Am J Hematol. Volume 93 Issue 3: pages 408-415, 2018 March).
FEV1/FVC Ratio Percentage | Through study completion, an average of four years
  Percentage of FEV1/FVC ratio based on the global lung index will be acquired from children with SCD receiving myeloablative curative therapies and adults with SCD receiving nonmyeloablative allo-HSCT, as well as from the respective control children and adult cohorts with SCD who received standard therapy. (References: Eur Respir J. Volume 40 Issue 6: pages 1324-1343, 2012 June 27; Am J Hematol. Volume 93 Issue 3: pages 408-415, 2018 March). FEV1/FVC will be reported in percentage.
Longitudinal change in eGFR | Through study completion, an average of four years
  Estimated GFR (eGFR) as a determinant of kidney disease will be collected from children with SCD receiving myeloablative curative therapies and adults with SCD receiving nonmyeloablative allo-HSCT, as well as from the respective control children and adult cohorts with SCD who received standard therapy. The eGFR will be tested as a linear variable and using eGFR Categories according to the KDIGO 2012 Guidelines (Table 5 - Reference: Kidney Int Suppl. Volume 3 Issue 1: pages 19-62, 2013 Jan) as follows:
  i.G1 >/ 90 mL/min/1.73m2 ii.G2 60 - 89 mL/min/1.73m2 iii.G3a 45 - 59 mL/min/1.73m2 iv.G3b 30 - 44 mL/min/1.73m2 v.G4 15 - 20 mL/min/1.73m2 vi.G5 < 15 mL/min/1.73m2 The standard technique of measured GFR will be used and reported in mL/min/1.73m2.
Longitudinal change in albuminuria levels | Through study completion, an average of four years
  Data pertaining to persistent albuminuria (defined as >/ 30 mg/g creatinine on 2 evaluations) associated with a more rapid decline in eGFR on longitudinal follow-up (Reference: Blood Adv. Volume 4 Issue 7: pages 1501-1511, 2020 Apr 14) will be tested. Results will be reported in mg/g.
Longitudinal change in TRJV in adults with SCD treated with nonmyeloablative allo HSCT in adults | Through study completion, an average of four years
  Improvement in TRJV in adults with SCD following HSCT will be acquired. Results will be reported in m/sec.
Longitudinal change in SBP/DBP in adults with SCD treated with nonmyeloablative allo HSCT in adults | Through study completion, an average of four years
  Measurements of Systolic blood pressure (SBP)/Diastolic blood pressure (DBP) in adults with SCD following HSCT will be acquired. Results will be reported as a ratio (SBP (mmHg)/DBP (mmHg)).

CONTACTS AND LOCATIONS:
Overall Officials: Michael R DeBaun, MD, MPH, Principal Investigator — Vanderbilt University Medical Center
Locations (5):
- United States (5):
  - Children's National Medical Center, Washington D.C., District of Columbia
  - Emory University School of Medicine, Atlanta, Georgia
  - Johns Hopkins Hospital, Baltimore, Maryland
  - National Institutes of Health Clinical Center, Bethesda, Maryland
  - Vanderbilt University Medical Center, Nashville, Tennessee

IPD SHARING:
Plan to Share IPD: Yes
This research study's sharing plan involves study data, publications, and outcomes. We will adhere to the NIH Public Access Policy (NOT-OD-08-033) and provide publications generated through funding by this project at the time the final, peer- reviewed papers are accepted for journal publication to the National Library of Medicine's PubMed Central, either through NIHMS (NIH Manuscript Submission) or through the Publisher. All applicable proposals, applications, and reports will include the PubMed Central number (PMCID) for all NIH-funded papers. All sequence data will be uploaded to database of Genotypes and Phenotype (dbGaP).